CLINICAL TRIAL: NCT03437603
Title: A Prospective Single-arm Study to Assess Efficacy and Safety of Eltrombopag For Secondary Poor Graft Function Post Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Eltrombopag For Secondary Poor Graft Function Post Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xiaowen Tang, Deputy director of Hematology Department，Clinical Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eltrombopag For PGF
Record Dates: First submitted 2018-01-27; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Poor Graft Function
Keywords: Eltrombopag; Allogenetic Hematopoietic Stem Cell Transplantation; Poor Graft Function
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag group (Experimental): Starting dose is 25mg daily for the first 3 days, then increasing to 50mg for another week. Maintenance dosage is 50mg or 75 mg per day dependent on patients' status and doctors' opinion.Planned duration of treatment with eltrombopag is 8 weeks.When patients achieve persistent complete response for 2 weeks,they may stop medicine.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Starting Eltrombopag daily on empty stomach (2 hour before breakfast) for 8 weeks.
  Other Names: Revolade

SUMMARY:
To investigate the efficacy and safety for secondary poor graft function (PGF) post allogeneic hematopoietic stem cell transplantation (allo-HSCT). The primary objective is the hematologic response rate. Secondary objectives include: (1) incidence and severity of adverse events; (2) overall survival (OS), and disease-free survival(DFS).

DETAILED DESCRIPTION:
Poor graft function (PGF) remains a life-threatening complication that occurs in 5-27% of patients following allogeneic hematopoietic stem cell transplantation (allo-HSCT), and is associated with morbidity and mortality related to infections or hemorrhagic complications.

PGF is defined below: (1) with two or three cytopenic lines (hemoglobin ≤70 g/L, neutrophil count ≤0.5×109/L, platelet count ≤20×109/L) with transfusion requirements; (2) with hypoplastic bone marrow and full donor chimerism; (3) without relapse or severe graft versus host diseases(GVHD) or active infectious diseases, or drug-related myelosuppression; (4) last at least for 14 conductive days. Primary PGF refers to those who did not achieve hematopoietic engraftment at day +28 post-transplant, while secondary PGF(sPGF)was defined as PGF after full engraftment.The underlying pathogenesis of PGF remains unclear. Therapeutic approaches for PGF include (1) growth factors, including granulocyte colony-stimulating factor (G-CSF), erythropoietin (EPO)- stimulating factors and thrombopoietin(TPO) mimetics; (2) second allo-HSCT; (3) infusion of additional mobilized cells from the original donor (modified DLI); (4) Cluster of differentiation 34（CD34）positive selected and T cell-depleted stem cell boost(SCB) without conditioning. and (5) mesenchymal stem cell(MSC) transfusion. However, second allo-HSCT and infusion of additional unmanipulated stem cells are associated with high rate of GVHD and treatment-related mortality (TRM). Up to now, there is no standard treatment recommended for PGF patients.

Eltrombopag is a kind of thrombopoietin receptor (TPO-R) agonists which can act as a stimulator of bone marrow progenitor cells.It has been approved by FDA for the treatment of immune thrombocytopenic purpura (ITP) and by European Union for severe aplasia anemia (SAA). Furthermore, there are also increasing amount of clinical trials using Eltrombopag for the treatment of thrombocytopenia post HSCT and very severe aplasia anemia(VSAA) which already had promising results. Due to the similarity in symptoms of PGF and AA, we suggested that if eltrombopag could be beneficial in patients with sPGF post allo-HSCT.

In this single-center open study,20 cases with sPGF post- transplant will be enrolled.The starting dose will be 25mg daily for 3 days to see if the drug is tolerable and then increasing to 50mg for another week. Maintenance dosage is 50mg or 75 mg per day dependent on patients' status and doctors' opinion.Patients may stop medicine when they achieve persistent complete response for 2 weeks.If patients only get partial response or no response after 8 weeks of therapy they may either stop eltrombopag or continue the drug considering doctor's advice. Once a patient suffer severe adverse events,patients should discontinue the drug immediately and get supporting measures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients develop poor graft function post allo-HSCT(primary or secondary),who had no response or were transfusion dependent after clinical therapeutic approaches(including growth factors,MSC transfusion,Cluster of differentiation(CD34) positive selected tem cell boosts infusion et al)
2. No recurrence or progression of primary malignancy after allo- HSCT
3. Patients with full donor chimerism
4. Patients without severe GVHD or active infectious diseases, or drug-related myelosuppression;
5. Written informed consent obtained from the subject.

Exclusion Criteria:

1. Alanine aminotransferase(ALT)≥2.5 times the upper limit of normal(ULN)
2. Serum bilirubin >2mg/dl
3. History of hepatic cirrhosis or the history of portal hypertension
4. Patients had any history of arterial / venous thrombosis within 1 year before enrollment in the study.
5. Take another treatment for drugs in 30 days or five half-life (no matter which longer) before the first drug delivery.
6. Eastern Cooperative Oncology Group(ECOG) performance status≥2.
7. Patients with a birth plan within 1 years, the pregnant or lactating women.
8. History of heart disease in the last 3 months, including congestive heart failure(III/IV Level, NHYA) ,arrhythmia, or myocardial infarction which medication is necessary. Any arrhythmia which could increase the risk of thrombotic events, or extended QT interval (QTc) of >480 milliseconds after correction.
9. Patients with cataract history；
10. Patients with myelofibrosis;
11. Patients who are unable to comply in the test and / or follow up stage.
12. Any abnormal situation in the screening stage or any other medical history or status that the researchers think is not suitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(Complete Response+Partial Response) | 8weeks
  Complete Response(CR)：CR was defined as neutrophil count ≥ 1.0×109/L independent of G-CSF for 3 consecutive days;platelets count ≥ 50×109/L without the need of platelet transfusion for at least 7 consecutive days;hemoglobin ≥ 90g/L.
  Partial response (PR)：Patients with at least 2 lines of blood cell count meeting the criteria of hematopoietic engraftment but not that of CR were defined as PR.

SECONDARY OUTCOMES:
Overall Survival(OS)/Disease Free Survival(DFS) | 12 months from study entry
  the survival rate after one year from study entry
Time to complete response | 8 weeks
  time when a patient achieve complete response
Time to achieve each lineage recovery | 8weeks
  time to achieve neutrophil/platelet/hemoglobin recovery respectively
Maintenance time after drug withdrawal | 12 months from study entry
  the recurrence time of poor graft function after drug withdrawal
Incidence of Adverse Events | 12months from study entry
  Safety profile Incidence of Adverse Events according to NCI Common Terminology Criteria for Adverse Events v 4.0 [NCI CTCAE] toxicity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, MD, Principal Investigator — The First Affliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China